CLINICAL TRIAL: NCT01285986
Title: Scandinavian Miller Collar Study
Acronym: SCAMICOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Sunderbyn Hospital (Other); Borås Lasarett (Other); Eskilstuna Lasarettet (Other); Falu Lasarett Röntgen (Other); Sahlgrenska University Hospital (Other); Lasarett Gävle (Other); Helsingborgs Hospital (Other); Kalmar County Hospital (Other); Karlstad Central Hospital (Other); Kristiansund Hospital (Other); Lund University Hospital (Other); Malmö University (Other); Department of Surgery, Lasarettet, Motala, Sweden (Unknown); Department of Surgery, Lasarettet, Mölndal, Sweden (Unknown); Department of Surgery, Lasarettet, Norrköping, Sweden (Unknown); Department of Surgery, Lasarettet, Nyköping, Sweden (Unknown); Department of Surgery, Lasarettet, Skellefteå, Sweden (Unknown); Department of Surgery, Kärnsjukhuset, Skövde, Sweden (Unknown); Department of Surgery, S:t Görans Sjukhus, Stockholm, Sweden (Unknown); Department of Surgery, Södersjukhuset, Stockholm, Sweden (Unknown); Department of Surgery, Norra Älvsborgs Länssjukhus, Trollhättan-Vänersborg, Sweden (Unknown); Uppsala University Hospital (Other); Västervik Hospital (Other); Region Västmanland (Other); Department of Surgery, Lasarettet, Växjö, Sweden (Unknown); Department of Surgery, Lasarettet, Örebro, Sweden (Unknown); Department of Surgery, Lasarettet, Östersund, Sweden (Unknown); Department of Vascular Surgery, Sykehuset, Kolding, Denmark (Unknown); Rigshospitalet, Denmark (Other); Aalborg University Hospital (Other)
Responsible Party: Fredrik Lundgren, Department od Cardiovascular Surgery, University Hospital, Linköping, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCAMICOS
Record Dates: First submitted 2011-01-27; First posted 2011-01-28 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Critical Limb Ischemia
Keywords: Graft patency; Limb salvage
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vein collar at distal anastomosis (Experimental): Vein collar at the distal anastomosis
  Interventions: Procedure: Vein collar at the distal anastomosis
- No vein collar at the distal anastomosis (Experimental): No vein collar at the distal anastomosis
  Interventions: Procedure: Vein collar at the distal anastomosis

INTERVENTIONS:
Procedure: Vein collar at the distal anastomosis — Vein collar interposed at the distal anastomosis or No vein collar interposed at the distal anastomosis

SUMMARY:
Randomized study to evaluate the effect of adding a vein collar at the distal anastomosis to PTFE-grafts used for bypass to below knee arteries in patients with critical limb ischemia with respect to primary patency, secondary patency, and limb salvage

ELIGIBILITY:
Inclusion Criteria:

* Critical limb ischemia
* Need for bypass surgery

Exclusion Criteria:

* Can not participate in follow-up
* Has suitable saphenous vein

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 1995-01; Primary Completion 1998-06 (Actual); Study Completion 1998-06 (Actual)

PRIMARY OUTCOMES:
Primary graft patency | Up to five years
  Follow-up at 1, 3, 6, and 12. Thereafter at most 5 years or until death of patient or amputation of limb. Primary graft patency = patent graft without any intervention to open up or prevent a graft ocklusion. Methods used for verification of patency: angiography, duplex, an improved ankle-brachial index was mantained, palpable pulse, or bi- or triphasic Doppler signal over the graft.

SECONDARY OUTCOMES:
Secondary Patency | Up to five years
  Secondary patency = patent graft after one or several interventions to open up or prevent a graft occlusion. Methods used for verification of secondary patency: angiography, duplex, an improved ankle-brachial index was mantained, palpable pulse, or bi- or triphasic Doppler signal over the graft.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik BG Lundgren, MD, PhD, Principal Investigator — Department of Cardiovascular Surgery, University Hospital, Linköping, Sweden
Locations (1):
- Department of CardioVascular Surgery, University Hospital, Linköping, Sweden